CLINICAL TRIAL: NCT03338673
Title: Neuromodulation Plus Cognitive Training to Improve Working Memory Among Individuals With Serious Mental Illness.
Brief Title: Brain Stimulation and Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Cynthia Burton, Clinical Lecturer, Department of Psychiatry, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HUM00119204
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Bipolar Disorder; Schizo Affective Disorder; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either dual therapy (cognitive exercises plus brain stimulation) or monotherapy (cognitive exercises alone) first; after 3 weeks participants will switch to the other condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Dual Therapy First (Experimental): Participants receive 10 sessions of non-invasive brain stimulation (tDCS) plus 10 hours of computerized cognitive exercises (BrainHQ), followed by 10 hours of computerized cognitive exercises alone
  Interventions: Device: tDCS; Other: BrainHQ
- Mono Therapy First (Experimental): Participants complete 10 hours of computerized cognitive exercises (BrainHQ) alone, followed by 10 sessions of non-invasive brain stimulation (tDCS) plus 10 hours of computerized cognitive exercises
  Interventions: Device: tDCS; Other: BrainHQ

INTERVENTIONS:
Device: tDCS — tDCS is a non-invasive procedure in which electrodes are attached to the scalp and send a small direct current to stimulate brain function
  Other Names: Transcranial direct current stimulation
Other: BrainHQ — BrainHQ is a web-based, commercially available cognitive training program that includes exercises to enhance working memory
  Other Names: Computerized cognitive exercises

SUMMARY:
People with serious mental illness often report difficulties with thinking skills like memory. These difficulties can make it harder to perform day-to-day activities. The purpose of this study is to test whether combining a type of non-invasive brain stimulation with computerized cognitive exercises is acceptable to participants, and whether it is helpful in improving a specific type of memory skill in people who have mental health conditions and memory deficits.

This study is designed so that all participants will get both treatments: the non-invasive brain stimulation and computerized cognitive exercises. Half of the participants will start with both the brain stimulation and the cognitive exercises (dual therapy), and half will start with just the computerized exercises (monotherapy). After three weeks, participants will switch to the other condition: the people who did both treatments first will switch to just the cognitive exercises alone, and the people who started with the cognitive exercises alone will then switch to doing both the brain stimulation and cognitive exercises.

Overall, participants will be in the study for about 7-8 weeks. The brain stimulation treatment involves 10 visits to the clinic over 3 weeks. The computerized cognitive exercises can be done at home, and involve 10 hours of exercises over 3 weeks. Participants will also complete paper-and-pencil assessments at the beginning, middle, and end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder I or II, schizoaffective disorder, or schizophrenia
* Objective cognitive impairment in working memory
* Willingness to complete computerized cognitive training and undergo brain stimulation procedures

Exclusion Criteria:

* History of neurological illness or brain injury (e.g., stroke)
* History of loss of consciousness
* Diagnosed intellectual disability
* Current substance use disorder
* Current mania or moderate depression or severe psychosis
* Serious suicidal ideation/behavior
* Pregnant or trying to become pregnant, or currently lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Burton, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dual Therapy First | Mono Therapy First
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dual Therapy First | Mono Therapy First | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.67 (13.98) | 48.83 (13.41) | 48.75 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participant Retention in Combination Treatment
Description: Number of participants completing every session of the combined phase of treatment
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dual Therapy First | Mono Therapy First
Number analyzed (Participants) | 6 | 6
Participants | 4 | 5

2. Primary Outcome: Participant-rated Acceptability of Combination Therapy
Description: Self-reported satisfaction as indicated on a numerical rating scale (1-10, where higher scores indicate greater satisfaction)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dual Therapy First | Mono Therapy First
Number analyzed (Participants) | 5 | 5
units on a scale | 9.40 (0.89) | 8.60 (2.07)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Dual Therapy First | Mono Therapy First
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03338673/Prot_SAP_000.pdf